CLINICAL TRIAL: NCT07340476
Title: A Phase I Study to Evaluate the PK Similarity of AK112 (Anti-PD-1/VEGF Bispecific Antibody) From the Proposed New Manufacturing Site and the Approved Original Site in Chinese Healthy Male Subjects.
Brief Title: A Study to Evaluate the PK Similarity of AK112 in Healthy Chinese Male Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AK112-105
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Healthy Male Subjects
Keywords: AK112

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK112 (New Site) (Experimental): AK112 (New Site) 3mg/kg, will be administrated intravenously in 60±10 minutes.
  Interventions: Drug: AK112 (New Site)
- AK112 (Original Site) (Active Comparator): AK112 (Original Site) 3mg/kg, will be administrated intravenously in 60±10 minutes.
  Interventions: Drug: AK112 (Original Site)

INTERVENTIONS:
Drug: AK112 (New Site) — AK112 (New Site) 3mg/kg
  Arms: AK112 (New Site)
Drug: AK112 (Original Site) — AK112 (Original Site)3mg/kg
  Arms: AK112 (Original Site)

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic (PK) similarity of AK112 (an anti-PD-1/VEGF bispecific antibody) from the proposed new manufacturing site and the approved original site in healthy male subjects.

Secondary objectives are to assess the safety, tolerability, and immunogenicity of AK112 from the proposed new manufacturing site and the approved original site.

ELIGIBILITY:
Inclusion Criteria:

1. Signing informed consent form before the trial and having a full understanding of the trial content, process and possible adverse reactions;
2. Able to complete the study according to the requirements of the study protocol.
3. Males aged 18 to 45;
4. Body Mass Index (BMI) is 19.0~26.0 kg/m2, and body weight is 55.0~75.0kg ;

Exclusion Criteria:

1. Those with a history of hypertension or blood pressure abnormalities at screening considered clinically significant by the investigator.
2. Those with a history of proteinuria or the presence of clinically significant proteinuria at screening as judged by the investigator.
3. Those with a history of severe bleeding tendency or coagulation dysfunction, or a history of thrombosis or hemorrhagic events; those with a history of esophageal-gastric varices, severe ulcers, gastrointestinal obstruction, or intra-abdominal abscess; those with a history of digestive tract perforation, hemorrhage, or fistula; those with a history of transient ischemic attack (TIA), cerebrovascular accident (stroke), hypertensive crisis, or hypertensive encephalopathy; those with a current unhealed wound or fracture.
4. Those with a history of autoimmune diseases (including personal or family history of hereditary immunodeficiency).
5. Those with a history of malignant tumor.
6. Those with a history of tuberculosis or clinical manifestations suspected to be tuberculosis (including but not limited to pulmonary tuberculosis, lymph node tuberculosis, tuberculous pleurisy, etc.).
7. Those with a history of recurrent or chronic infections, including a history of chronic or recurrent infections such as: chronic kidney infection, chronic thoracic cavity infection (e.g., bronchiectasis), sinusitis, recurrent urinary tract infections, open, draining, or infected skin wounds.
8. Those with a history of acute infection within 4 weeks prior to randomization; or those with a history of opportunistic infections (e.g., herpes zoster, active cytomegalovirus, Pneumocystis jirovecii, histoplasmosis, aspergillosis, mycobacterial infections, etc.) within 6 months prior to randomization.
9. Those who underwent major surgery within 3 months prior to randomization or experienced serious trauma, or those who plan to undergo surgical procedures during the trial period.
10. Those who donated blood or experienced significant blood loss (≥400 mL) within 3 months prior to randomization, received blood transfusion or blood products, or plan to donate blood or blood components during the trial period or within 3 months after completion of the trial.
11. Those unable to tolerate venipuncture or with a history of fainting during blood draws or injections (vasovagal reaction).
12. Those with a known allergy to any component of the investigational product, or those with a history of allergy to two or more drugs, foods, or other substances.
13. Those with a history of other diseases affecting the digestive, respiratory, cardiovascular, endocrine, urinary, neurological, hematologic, or metabolic systems that the investigator deems to have ongoing clinical significance.
14. Those with a positive result in the urine drug screen test (for morphine, methamphetamine, ketamine, methylenedioxymethamphetamine [MDMA], tetrahydrocannabinol [THC]).
15. Those with a positive alcohol breath test.
16. Those who test positive for any of the following: Human Immunodeficiency Virus (HIV) antibody, Hepatitis C Virus (HCV) antibody, Syphilis test (RPR), Hepatitis B Virus (HBV) surface antigen, e-antigen (HBeAg), or core antibody (HBcAb).
17. Those with abnormal findings in other examinations (physical examination, vital signs, chest X-ray, laboratory tests, etc.) that are considered clinically significant by the investigator.
18. Those who have previously used any drug targeting PD-1, PD-L1, VEGF, or VEGFR pathways.
19. Those who received other investigational medicinal products or participated in another interventional clinical trial within 3 months prior to randomization.
20. Those vaccinated with live or attenuated vaccines within 3 months prior to randomization, or those vaccinated with inactivated vaccines within 14 days prior to randomization, or those who plan to receive vaccinations during the trial period.
21. Those who used any medication (including traditional Chinese medicine, health supplements, etc.) within 14 days prior to randomization, or those whose last dose was administered less than 5 half-lives before the randomization date, whichever is longer.
22. Those with a history of drug abuse or those who used soft drugs (e.g., marijuana) or hard drugs (e.g., cocaine, phencyclidine, etc.) within 1 year prior to receiving the investigational product.
23. Those who are smokers or smoked more than 5 cigarettes per day within 3 months prior to randomization, or those unable to abstain from all tobacco products during hospitalization.
24. Those who are heavy drinkers or frequent drinkers within 12 months prior to randomization, defined as consuming more than 14 units of alcohol per week (1 unit = 360 mL beer or 45 mL spirits [40% alcohol] or 150 mL wine); or those unwilling to abstain from alcohol or any alcoholic beverages during the trial period.
25. Those with special dietary requirements that prevent compliance with the standardized diet, or those who are lactose intolerant.
26. Those whose subject or partner has plans for pregnancy during the study period through 3 months after trial completion, or those unwilling to use reliable contraceptive measures (such as abstinence, sterilization, oral contraceptives, injectable contraceptives like medroxyprogesterone acetate, subdermal implants, condoms, etc.).
27. Those who may be unable to complete this study for other reasons, or those unable to comply with the study procedures during the study period, or those deemed by the investigator to have other reasons making them unsuitable for participation in the trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is based on biological sex and reproductive risk criteria; gender identity is not a basis for exclusion.
Enrollment: 108 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC0-infinity) | From pre-dose to day 43

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC0-t) | From pre-dose to day 43
Maximum plasma concentration (Cmax) | From pre-dose to day 43
Volume of distribution (Vd) | From pre-dose to day 43
Clearance (CL) | From pre-dose to day 43
Ratio of AUC0-t/AUC0-infinity | From pre-dose to day 43
Time to maximum concentration (Tmax) | From pre-dose to day 43
Half-life (t1/2) | From pre-dose to day 43
Incidence and severity of adverse events (AEs) | Up to day 43
Number and percentage of subjects with detectable ADA | From pre-dose to day 43

CONTACTS AND LOCATIONS:
Overall Officials: Jinliang Chen, MD, Principal Investigator — Zhejiang Hospital
Locations (1):
- Zhejiang Xiaoshan Hospital, Zhejiang, Xiaoshan, China